CLINICAL TRIAL: NCT03346616
Title: Text4Peds: Randomized Controlled Trial Evaluating Medical Student Education
Brief Title: Text4Peds: Short Message Service Evaluating Medical Student Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Matthew A. Broom, MD, FAAP, Associate Professor of Pediatrics, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 26458
Record Dates: First submitted 2017-10-30; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Education, Medical, Undergraduate; SMS

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to a Texting Group or a Non-Texting Group using a random number generator. The texting group received a daily text message containing a board style multiple choice question. If the participant wanted immediate feedback, the message contained a link to a website containing the answer to the question along with an explanation, the source material, and a more complete clinical vignette. One hour after the initial text message was sent, a follow up "answer" text message was delivered. Text messages were sent 6 days per week (Monday through Saturday) at 2pm and 3pm. To minimize perceived impropriety, the non-texting group received access to the journal articles from which the content was derived, but did not receive any text messages or any of the synthesized material. The primary outcome was performance on the NBME Pediatric Subject Examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Texting Group (Experimental): The texting group received a daily text message containing a board style multiple choice question. If the participant wanted immediate feedback, the message contained a link to a website containing the answer to the question along with an explanation, the source material, and a more complete clinical vignette. One hour after the initial text message was sent, a follow up "answer" text message was delivered. Text messages were sent 6 days per week (Monday through Saturday) at 2 pm and 3 pm.
  Interventions: Other: Texting Group
- Non Texting Group (Active Comparator): The non-texting group received access to the journal articles from which the text message content was derived, but did not receive any text messages or any of the online material or question stems.
  Interventions: Other: Non Texting Group

INTERVENTIONS:
Other: Texting Group — See above in arm/group description
  Arms: Texting Group
Other: Non Texting Group — See above in arm/group description
  Arms: Non Texting Group

SUMMARY:
In this study, third year medical students on the pediatric clerkship will be randomized to receive either only written educational material (review journal articles) or written educational material plus daily text messages consisting of board style questions with online answers. The students' performance on the National Board of Medical Examiners (NBME) Pediatric Subject Evaluation will be compared between the two groups.

DETAILED DESCRIPTION:
In the last decade, the use of smartphone and text messaging (SMS) has increased significantly; during this time, text messaging has become the primary means of communication in some instances. Despite the popularity, text messaging and smartphones have been rarely utilized in the context of medical education. Few studies have been performed examining the effect of text messaging as an adjunct to traditional medical education. A previous study with the Saint Louis University (SLU) Pediatric Residency program, showed the feasibility of using text messaging to deliver medical information to pediatric residents through the Text4Peds program.

This study aims to expand Text4Peds to third NBME Pediatric Subject Evaluation performance. The NBME Pediatric Subject Evaluation is a national, standardized pediatric knowledge based exam from the NBME taken by all medical students at the end of their pediatric clerkship.

ELIGIBILITY:
Inclusion Criteria:

* Third year medical students on the Pediatric Clerkship at Saint Louis University School of Medicine

Exclusion Criteria:

* Third year medical students who did not have a mobile phone capable of receiving a short message service (SMS) text message

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
National Board of Medical Examiners Pediatric Subject Examination | Assessed at end of intervention (after 8 weeks)
  The NBME pediatrics subject examination is used to assess medical student knowledge and is a common component of the pediatric clerkship grade. It is also used to compare medical student performance to a national benchmark. NBME scores are on a scale of 0-100 (% correct); mean score for this exam during year of evaluation was 75.7 (SD 8.7).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Brownsworth, MD, Principal Investigator — St. Louis University
Locations (1):
- St Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gavali MY, Khismatrao DS, Gavali YV, Patil KB. Smartphone, the New Learning Aid amongst Medical Students. J Clin Diagn Res. 2017 May;11(5):JC05-JC08. doi: 10.7860/JCDR/2017/20948.9826. Epub 2017 May 1. PMID 28658804
- [Background] Stockwell MS, Kharbanda EO, Martinez RA, Lara M, Vawdrey D, Natarajan K, Rickert VI. Text4Health: impact of text message reminder-recalls for pediatric and adolescent immunizations. Am J Public Health. 2012 Feb;102(2):e15-21. doi: 10.2105/AJPH.2011.300331. Epub 2011 Dec 15. PMID 22390457
- [Background] Goodarzi M, Ebrahimzadeh I, Rabi A, Saedipoor B, Jafarabadi MA. Impact of distance education via mobile phone text messaging on knowledge, attitude, practice and self efficacy of patients with type 2 diabetes mellitus in Iran. J Diabetes Metab Disord. 2012 Aug 31;11(1):10. doi: 10.1186/2251-6581-11-10. PMID 23497632
- [Background] Hall AK, Cole-Lewis H, Bernhardt JM. Mobile text messaging for health: a systematic review of reviews. Annu Rev Public Health. 2015 Mar 18;36:393-415. doi: 10.1146/annurev-publhealth-031914-122855. PMID 25785892
- [Background] Sabin LL, Larson Williams A, Le BN, Herman AR, Viet Nguyen H, Albanese RR, Xiong W, Shobiye HO, Halim N, Tran LTN, McNabb M, Hoang H, Falconer A, Nguyen TTT, Gill CJ. Benefits and Limitations of Text Messages to Stimulate Higher Learning Among Community Providers: Participants' Views of an mHealth Intervention to Support Continuing Medical Education in Vietnam. Glob Health Sci Pract. 2017 Jun 27;5(2):261-273. doi: 10.9745/GHSP-D-16-00348. Print 2017 Jun 27. PMID 28655802
- [Background] Gill CJ, Le Ngoc B, Halim N, Nguyen Viet H, Larson Williams A, Nguyen Van T, McNabb M, Tran Thi Ngoc L, Falconer A, An Phan Ha H, Rohr J, Hoang H, Michiel J, Nguyen Thi Thanh T, Bird L, Pham Vu H, Yeshitla M, Ha Van N, Sabin L. The mCME Project: A Randomized Controlled Trial of an SMS-Based Continuing Medical Education Intervention for Improving Medical Knowledge among Vietnamese Community Based Physicians' Assistants. PLoS One. 2016 Nov 18;11(11):e0166293. doi: 10.1371/journal.pone.0166293. eCollection 2016. PMID 27861516
- [Background] Chen Y, Yang K, Jing T, Tian J, Shen X, Xie C, Ma B, Liu Y, Yao L, Cao X. Use of text messages to communicate clinical recommendations to health workers in rural China: a cluster-randomized trial. Bull World Health Organ. 2014 Jul 1;92(7):474-81. doi: 10.2471/BLT.13.127076. Epub 2014 Mar 25. PMID 25110372
- [Background] Gurol-Urganci I, de Jongh T, Vodopivec-Jamsek V, Atun R, Car J. Mobile phone messaging reminders for attendance at healthcare appointments. Cochrane Database Syst Rev. 2013 Dec 5;2013(12):CD007458. doi: 10.1002/14651858.CD007458.pub3. PMID 24310741
- [Background] Mount HR, Zakrajsek T, Huffman M, Deffenbacher B, Gallagher K, Skinker B, Rivard G, Benson S, Dancel R, Buckman F, Hayes M, Jackson J, Viera AJ. Text messaging to improve resident knowledge: a randomized controlled trial. Fam Med. 2015 Jan;47(1):37-42. PMID 25646876
- [Background] Draper L, Kuklinski C, Ladley A, Adamson G, Broom M. Texting preferences in a Paediatric residency. Clin Teach. 2017 Dec;14(6):401-406. doi: 10.1111/tct.12590. Epub 2017 Jan 12. PMID 28078778
- [Background] Broom MA, Adamson GT, Draper LR. Text messaging in medical education. Pediatrics. 2014 Mar;133(3):e491-3. doi: 10.1542/peds.2013-1529. Epub 2014 Feb 17. No abstract available. PMID 24534409

DOCUMENTS (3):
  • Study Protocol (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03346616/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03346616/SAP_001.pdf
  • Informed Consent Form (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03346616/ICF_002.pdf